CLINICAL TRIAL: NCT03804775
Title: Comparative Analysis of Serum Lipid Profiles in Patients With and Without Gallstones: A Prospective Cross-Sectional Study
Brief Title: Comparative Analysis of Serum Lipid Profiles in Patients With and Without Gallstones
Status: Completed | Type: Observational
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Other Study IDs: s10
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Gallstone; Dyslipidemias
MeSH Terms: conditions — Gallstones; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: patients presenting with gallstone disease
  Interventions: Diagnostic Test: Serum lipid profile
- control group: inpatients with no history of gallstones
  Interventions: Diagnostic Test: Serum lipid profile

INTERVENTIONS:
Diagnostic Test: Serum lipid profile — Blood samples drawn from the patients and controls will be analyzed for serum cholesterol, serum triglycerides, serum LDLs and serum HDL levels. All the results will be recorded on a performa

SUMMARY:
Gallbladder disease is one of the most common diseases of the gastrointestinal tract. Various studies have shown an association between gallstones and an alteration in the serum lipids. The objective of this study will be to compare serum lipid profile of gallstone patients with the controls.

DETAILED DESCRIPTION:
This prospective cross-sectional study will be conducted in the Surgical Department of the Services Institute of Medical Sciences. A total of 50 patients will beincluded in the study after screening through the inclusion criteria. A control group of 50 inpatients with no personal or family history of gallstones will be also recruited for comparison. Results will be expressed as mean with standard deviation. Students t- test will be used to compare the data between the patients and the control groups (p<0.05 will be considered statistically significant). SPSS software, version 20 will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with the gall stone disease
* Age from 20 to 70 years
* Gallstones were diagnosed through the ultrasound

Exclusion Criteria:

* Patients with acalculous gallbladder disease on ultrasound,
* Patients with terminal ileal resection,
* Patients with hemolytic diseases (hereditary spherocytosis, sickle cell anemia on history and CBC film),
* Patients with liver cirrhosis (on abdominal ultrasound) and
* Patients on antihyperlipidemic drugs

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Case group: patients from lahore city presented with gallstone disease in Services Hospital lahore
  Control group: Patients admitted to Services Hospital with other diseases belonging from lahore
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
serum cholesterol levels | 1 week
  serum cholesterol levels of patients and case group will be compared with Students t- test was (p<0.05 will be considered statistically significant)
serum triglyceride levels | 1 week
  serum triglyceride levels of gallstone patients and control group will be compared via student t-test (p<0.05 was considered statistically significant)
serum HDL levels | 1 week
  serum HDL levels of patients and contoled will be compared with student t-test (p<0.05 was considered statistically significant)
serum LDL leves | 1 week
  serum LDL leves of patients and control will be compared through student t-test (p<0.05 was considered statistically significant)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided